CLINICAL TRIAL: NCT01578421
Title: Investigation on the Middle Size Molecule Elimination Characteristics of the FXCorDiax 100 in Relation to the FX 100 and the Polyflux 210 H Dialyser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Aarau (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Principal Investigator, Andreas Bock, Prof. Andreas Bock, Chefarzt Nephrologie, Kantonsspital Aarau
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD-FX-01-CH
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FX 100 dialyzer (Other)
  Interventions: Device: 4 h online hemodiafiltration (FX 100, Polyflux 210, FXCorDiax)
- Polyflux 210 H dialyzer (Other)
  Interventions: Device: 4 h online hemodiafiltration (FX 100, Polyflux 210, FXCorDiax)
- FXCorDiax 100 dialyzer (Other)
  Interventions: Device: 4 h online hemodiafiltration (FX 100, Polyflux 210, FXCorDiax)

INTERVENTIONS:
Device: 4 h online hemodiafiltration (FX 100, Polyflux 210, FXCorDiax) — 4 h online hemodiafiltration with measurement of clearance and removal rate by split dialysate collection and bloodside measurements

SUMMARY:
The purpose of the study is to compare clearance and removal rates of phosphate, ß2-microglobulin (ß2-m) and leptin and albumin loss with different dialyser membranes during post-dilution online hemodiafiltration.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients 18 years and older
* treated by post dilution on-line Hemodiafiltration (HDF) for at least one month
* who reached a dialysis dose (Kt/V) of at least 1.2 at each of the last two monthly checks
* who are on a stable anticoagulation and anemia management
* whose hemoglobin is between 10.5 and 13.0 g/dl
* who are clinically stable based on judgment of nephrologist
* who are on a regular thrice weekly HDF schedule, e.g. Monday-Wednesday-Friday or Tuesday-Thursday-Saturday,
* who have a good vascular access (fistula or graft) which enables easy insertion of the needles and suitable effective blood flow (> 300 ml/min)
* who are able to understand the nature and requirements of the clinical investigation and who have given written informed consent

Exclusion Criteria: Patients

* with active Hepatitis B, Hepatitis C or HIV infection
* who are severely malnourished as judged by the principal investigator
* who are known or suspected to have allergy to the trial products or related products
* with a central venous catheter based vascular access
* who are abusing non-legal drugs or alcohol
* who have currently active malignant disease
* who are female of child-bearing age without effective measures of contraception, pregnant or breastfeeding
* who participate simultaneously in another clinical investigation
* who have participated in othe clinical investigations during the last month
* who are uncooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Clearance and removal rate of phosphate, beta2 microglobulin and leptin | 4 hour
  during a 4 hour online hemodiafiltration session

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bock, MD, Principal Investigator — Nephrology Division, Kantonsspital Aarau
Locations (1):
- Nephrology Division, Kantonsspital Aarau, Aarau, Switzerland